CLINICAL TRIAL: NCT05926102
Title: The Prostate Cancer, Genetic Risk, and Equitable Screening Study (ProGRESS): A Pragmatic Trial of Precision Prostate Cancer Screening
Brief Title: The Prostate Cancer, Genetic Risk, and Equitable Screening Study (ProGRESS)
Acronym: ProGRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ONCA-021-22F; I01CX002635 (NIH)
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: early detection of cancer; prostatic neoplasms; polygenic risk scores; family health history
MeSH Terms: conditions — Prostatic Neoplasms; Genetic Risk Score

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomly allocated to receive either the precision screening intervention or usual care. The precision screening intervention will consist of an interpreted prostate cancer genetic risk assessment (GRA) report, provided to the participant along with tailored prostate cancer screening recommendations and, in cases of high genetic risk, genetic counseling. The risk report and supporting educational materials will also be provided to the participant's primary care provider. Usual care in this study includes receipt of a brief brochure about shared decision-making in prostate cancer screening.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Precision screening intervention (Experimental): The precision screening intervention will consist of an interpreted prostate cancer genetic risk assessment (GRA) report, provided to the participant along with tailored prostate cancer screening recommendations and, in cases of high genetic risk, genetic counseling. The risk report and supporting educational materials will also be provided to the participant's primary care provider. Usual care in this study includes receipt of a brief brochure about shared decision-making in prostate cancer screening.
  Interventions: Genetic: Precision screening intervention; Other: Usual care
- Usual care (Experimental): Usual care in this study includes receipt of a brief brochure about shared decision-making in prostate cancer screening.
  Interventions: Other: Usual care

INTERVENTIONS:
Genetic: Precision screening intervention — The precision screening intervention will consist of an interpreted prostate cancer genetic risk assessment (GRA) report, provided to the participant along with tailored prostate cancer screening recommendations and, in cases of high genetic risk, genetic counseling. The risk report and supporting educational materials will also be provided to the participant's primary care provider. Usual care in this study includes receipt of a brief brochure about shared decision-making in prostate cancer screening.
  Arms: Precision screening intervention
Other: Usual care — Usual care in this study includes receipt of a brief brochure about shared decision-making in prostate cancer screening.

SUMMARY:
Prostate cancer is the most common non-skin cancer among Veterans and the second leading cause of male cancer death. Current methods of screening men for prostate cancer are inaccurate and cannot identify which men do not have prostate cancer or have low-grade cases that will not cause harm and which men have significant prostate cancer needing treatment. False-positive screening tests can result in unnecessary prostate biopsies for men who do not need them. However, new genetic testing might help identify which men are at highest risk for prostate cancer. This study will examine whether a genetic test helps identify men at risk for significant prostate cancer while helping men who are at low risk for prostate cancer avoid unnecessary biopsies. If this genetic test proves beneficial, it will improve the way that healthcare providers screen male Veterans for prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-cutaneous cancer in US men and in the Veterans Health Administration (VHA): 1 in 8 will be diagnosed with the disease in their lifetime. Many cases are non-lethal, but prostate cancer remains the 2nd leading cause of cancer death among US men, representing 2.5% of all deaths. VHA diagnoses >16,000 new cases annually and cares for >400,000 men living with prostate cancer. As a result, prostate cancer diagnosis and treatment is a national priority for VHA.

A major impediment to reducing the incidence of metastatic prostate cancer and prostate cancer death is the lack of an optimal screening strategy to identify men at high risk. Screening with prostate-specific antigen (PSA) testing modestly reduces prostate cancer deaths but at the cost of overdiagnoses and overtreatment. Current screening approaches do not adequately distinguish men without prostate cancer or with low-grade prostate cancer amenable to active surveillance from men with clinically significant prostate cancer, who need treatment. As a result, clinical guidelines do not recommend universal prostate cancer screening, including those from the United States Preventive Services Task Force (USPSTF) and the VHA National Center for Health Promotion and Disease Prevention. Still, many men undergo screening based on variable and subjective assessments of their race/ethnicity, family history, and other risk factors.

A new paradigm of precision screening could improve the benefit-to-harm ratio of screening by implementing screening strategies tailored to an individual's specific genetic profile. Due to advances in high-throughput genotyping and sequencing, increasingly large and diverse cohort studies, and standardization of genetic variant classification, germline genetic testing is emerging as a powerful predictor for prostate cancer, including metastatic and lethal disease. This includes both rare highly penetrant variants and polygenic risk scores (PRS), which characterize an individual's predisposition to prostate cancer due to common genetic variation. Rare and common genetic variation is now an equally powerful predictor of clinically significant disease as self-reported race or family history, including in the Million Veteran Program.

This clinical trial will evaluate the promise of precision risk stratification to identify men most likely to benefit from prostate cancer screening. During the proof-of-concept phase, the investigators will achieve the following aims:

1. Develop a precision prostate cancer screening intervention consisting of genetic testing for rare variants and a transancestry PRS, delivered to participants and their primary care providers along with individualized, genetic risk-informed screening recommendations.
2. Determine the feasibility of enrolling men aged 55-70 ( 35% of whom are of racial/ethnic minority groups) to a pragmatic randomized clinical trial (RCT) comparing the precision screening intervention to usual care.
3. Perform an interim assessment to determine whether the observed trajectory of negative prostate biopsy event rates is consistent with rates needed to detect a meaningful between-group difference at the end of the 7-year project period.

If the investigators demonstrate feasibility of enrollment and adequate event rates during the proof-of-concept phase, the RCT will continue to the clinical trial phase to test the following co-primary hypotheses:

1. Compared with men in the usual care arm, men in the precision screening arm will have a time-to-diagnosis of clinically significant prostate cancer (csPCa, defined as NCCN classification intermediate risk or higher) that is not inferior by a margin of >30 days over a median 4 years of follow-up.

   a. If non-inferiority is demonstrated, the investigators will sequentially test the hypothesis that time-to-diagnosis of csPCa is shorter in the precision screening arm than in the usual care arm (superiority).
2. Compared with usual care, men in the precision screening arm overall will undergo fewer negative prostate biopsies over a median 4 years of follow-up.

Pre-specified subgroup analyses will test these hypotheses in Black men specifically, to evaluate whether this population benefits equally or more from the intervention. Enrollees will be followed for additional outcomes including all prostate cancer diagnoses, PSA testing, prostate MRI, rare variants identified, preferences for or against prostate cancer screening, and health-related quality of life.

The investigators expect that precision screening will increase screening among high-risk patients but decrease screening among low- and average-risk patients, thereby maintaining or improving overall csPCa detection while improving the population-level benefit-to-harm ratio. Rigorous RCT evidence that genetic risk-informed screening maintains the benefits of screening while minimizing the harms of unnecessary procedures and treatments among low-risk men will change clinical practice and policy around prostate cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* baseline age 55-69 years
* receipt of regular VA care
* Veteran status

Exclusion Criteria:

* personal history of prostate cancer
* prior prostate biopsy, prostatectomy, or prostate MRI
* known carrier status of rare variant associated with cancer syndrome

Ages: 55 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of clinically significant prostate cancer | 7 years
  Cases of csPCa will be abstracted from VA and survey data and defined using NCCN classifications of intermediate risk or higher: PSA 10 and/or Grade Group 2 and/or clinical T stage T2b
Negative prostate biopsy | 7 years
  Counts of negative prostate biopsies not temporally associated with csPCa (within 6 months of diagnosis) will be abstracted from VA and survey data

SECONDARY OUTCOMES:
Diagnosis of prostate cancer | 7 years
  All cases of prostate cancer will be abstracted from VA and survey data
Prostate biopsy | 7 years
  Counts of all prostate biopsies will be abstracted from VA and survey data.
PSA testing | 7 years
  PSA testing will be identified from VA and survey data
Prostate MRI | 7 years
  Prostate magnetic resonance imaging will be identified from VA and survey data
Self-rated health | 7 years
  Self-rated health will be collected at the baseline survey and every 6 months with a single-item self-rating of health on a Likert scale from "poor" to "excellent.
Quality of life | 5 years
  Health-related quality of life is collected through the Veterans RAND 12-Item Health Survey (VR-12) on the baseline survey and at each participant's 5-year survey or last survey

OTHER OUTCOMES:
Adherence to precision cancer screening recommendations | 7 years
  The precision screening intervention will include the recommendation that high-risk men undergo PSA screening and that low-risk men not undergo screening. The investigators will define adherence to the intervention in these two groups of men as the presence and absence of PSA testing, respectively, during the observation period.
Acceptability of the precision prostate cancer screening intervention | 7 years
  The survey will assess patient acceptability of the precision screening with a 3-item instrument assessing patient perspective on the 1) amount of information presented, 2) length of the information, 3) clarity of the information, with each domain scored on a 5-point Likert scale.
Rare pathogenic/likely pathogenic variants | 7 years
  Proportion of participants with a rare P/LP variant associated with hereditary prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Vassy, MD MPH, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be stored in a data repository available for request by approved individuals.
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: Requestors may be required to have IRB approval, data use agreements, and other regulatory and administrative credentials and authorizations prior to receiving data.

REFERENCES:
- [Derived] Vassy JL, Dornisch AM, Karunamuni R, Gatzen M, Kachulis CJ, Lennon NJ, Brunette CA, Danowski ME, Hauger RL, Garraway IP, Kibel AS, Lee KM, Lynch JA, Maxwell KN, Ratner D, Rose BS, Teerlink CC, Xu GJ, Hofherr SE, Lafferty KA, Larkin K, Malolepsza E, Patterson CJ, Toledo DM, Donovan JL, Hamdy FC, Martin RM, Neal DE, Turner EL, Andreassen OA, Dale AM, Mills IG, Abraham A, Batra J, Clements J, Cussenot O, Cybulski C, Eeles RA, Fowke JH, Grindedal EM, Gronberg H, Hamilton RJ, Lim J, Lu YJ, MacInnis RJ, Maier C, Mucci LA, Multigner L, Neuhausen SL, Nielsen SF, Parent ME, Park JY, Petrovics G, Plym A, Razack A, Rosenstein BS, Schleutker J, Sorensen KD, Townsend PA, Travis RC, Vega A, West CML, Wiklund F, Zheng W; Profile Steering Committee; IMPACT Study Steering Committee and Collaborators; PRACTICAL Consortium; VA Million Veteran Program; Seibert TM. Genomic risk model to implement precision prostate cancer screening in clinical care: the ProGRESS study. Nat Cancer. 2026 Jan 26. doi: 10.1038/s43018-025-01103-0. Online ahead of print. PMID 41588240